CLINICAL TRIAL: NCT00022750
Title: Project Sugar 2: Health Events Costs in Diabetic Blacks
Brief Title: Randomized Trial of Health Events Costs in Diabetic Blacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: DK48117 (completed); R01DK048117-06 (NIH); OPD-GCRC R00052
Record Dates: First submitted 2001-08-10; First posted 2001-08-10 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; Nurse Case Manager; Community Health Worker; Behavioral Interventions; Cost-effectiveness; Randomized trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: Nurse Case Manager and Community Health Worker Team

SUMMARY:
Diabetes mellitus imposes a major burden on the public health of the United States, leading annually to over 300,000 deaths and over $130 billion in costs. This burden falls disproportionately upon ethnic minority groups, particularly African Americans, who are at excess risk for the development of type 2 diabetes and for a variety of its most serious complications. Suboptimal health care - in terms of access, quality, and adherence -appears to be an important contributing factor. Prior work suggests two possible approaches aimed at prevention to enhance risk factor control in outpatients with type 2 diabetes. One approach uses Nurse Case Managers (NCMs) to coordinate care plans with the provider team following protocols/clinical guidelines and algorithms designed to guide treatment including initiating and adjusting drug therapy, enhancing continuity of care, promoting interventions and self-management which include educational and behavioral strategies incorporating feedback and self-regulation. Another approach uses Community Health Workers (CHWs) to enhance culturally sensitive outreach, linkage, and monitoring service; to provide important patient and family education; and to improve access to and continuity of care. Results indicate that this intensive team approach, compared to usual care alone, produces substantial improvements in metabolic control. However, the cost-effectiveness of such interventions is unknown in the ''real-world''.

This has led to our current study, a randomized controlled trial within a managed care organization to determine the effects of a NCM/CHW team on metabolic control, on the occurrence of diabetes-related health events, health care utilization, and on direct health care costs. The participants will be African American adults with type 2 diabetes who receive primary care within a managed care organization in inner-city Baltimore.

ELIGIBILITY:
Inclusion Criteria:

* African American male or female aged 30 years or older diagnosed with type 2 diabetes mellitus
* Able to provide 2 contact persons outside his/her household with active, verified telephone numbers

Exclusion Criteria:

* Mentally incompetent to give informed consent
* Refuses to give informed consent
* Comorbid health condition likely to lead to death in next 24 months

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2000-10; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L. Brancati, MD, MHS, Principal Investigator — The Johns Hopkins Medical Institutions
Locations (1):
- The Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

REFERENCES:
- [Background] Brancati FL, Whittle JC, Whelton PK, Seidler AJ, Klag MJ. The excess incidence of diabetic end-stage renal disease among blacks. A population-based study of potential explanatory factors. JAMA. 1992 Dec 2;268(21):3079-84. PMID 1433738
- [Background] Brancati FL, Appel LJ, Seidler AJ, Whelton PK. Effect of potassium supplementation on blood pressure in African Americans on a low-potassium diet. A randomized, double-blind, placebo-controlled trial. Arch Intern Med. 1996 Jan 8;156(1):61-7. PMID 8526698
- [Background] Krop JS, Coresh J, Chambless LE, Shahar E, Watson RL, Szklo M, Brancati FL. A community-based study of explanatory factors for the excess risk for early renal function decline in blacks vs whites with diabetes: the Atherosclerosis Risk in Communities study. Arch Intern Med. 1999 Aug 9-23;159(15):1777-83. doi: 10.1001/archinte.159.15.1777. PMID 10448782
- [Background] Hill MN, Becker DM. Roles of nurses and health workers in cardiovascular health promotion. Am J Med Sci. 1995 Dec;310 Suppl 1:S123-6. doi: 10.1097/00000441-199512000-00022. PMID 7503115
- [Background] Shediac-Rizkallah MC, Bone LR. Planning for the sustainability of community-based health programs: conceptual frameworks and future directions for research, practice and policy. Health Educ Res. 1998 Mar;13(1):87-108. doi: 10.1093/her/13.1.87. PMID 10178339
- [Background] Levine DM, Becker DM, Bone LR, Hill MN, Tuggle MB 2nd, Zeger SL. Community-academic health center partnerships for underserved minority populations. One solution to a national crisis. JAMA. 1994 Jul 27;272(4):309-11. No abstract available. PMID 8028145
- [Background] Krop JS, Powe NR, Weller WE, Shaffer TJ, Saudek CD, Anderson GF. Patterns of expenditures and use of services among older adults with diabetes. Implications for the transition to capitated managed care. Diabetes Care. 1998 May;21(5):747-52. doi: 10.2337/diacare.21.5.747. PMID 9589235
- [Background] Powe NR, Weiner JP, Starfield B, Stuart M, Baker A, Steinwachs DM. Systemwide provider performance in a Medicaid program. Profiling the care of patients with chronic illnesses. Med Care. 1996 Aug;34(8):798-810. doi: 10.1097/00005650-199608000-00007. PMID 8709661
- [Result] Hill-Briggs F, Gary TL, Yeh HC, Batts-Turner M, Powe NR, Saudek CD, Brancati FL. Association of social problem solving with glycemic control in a sample of urban African Americans with type 2 diabetes. J Behav Med. 2006 Feb;29(1):69-78. doi: 10.1007/s10865-005-9037-0. Epub 2006 Jan 6. PMID 16397820
- [Result] Jackson CL, Bolen S, Brancati FL, Batts-Turner ML, Gary TL. A systematic review of interactive computer-assisted technology in diabetes care. Interactive information technology in diabetes care. J Gen Intern Med. 2006 Feb;21(2):105-10. doi: 10.1111/j.1525-1497.2005.00310.x. Epub 2005 Dec 22. PMID 16390512
- [Result] Gary TL, Maiese EM, Batts-Turner M, Wang NY, Brancati FL. Patient satisfaction, preventive services, and emergency room use among African-Americans with type 2 diabetes. Dis Manag. 2005 Dec;8(6):361-71. doi: 10.1089/dis.2005.8.361. PMID 16351554
- [Result] Gary TL, Hill-Briggs F, Batts-Turner M, Brancati FL. Translational research principles of an effectiveness trial for diabetes care in an urban African American population. Diabetes Educ. 2005 Nov-Dec;31(6):880-9. doi: 10.1177/0145721705282254. PMID 16288095
- [Result] Jackson CL, Batts-Turner ML, Falb MD, Yeh HC, Brancati FL, Gary TL. Computer and internet use among urban African Americans with type 2 diabetes. J Urban Health. 2005 Dec;82(4):575-83. doi: 10.1093/jurban/jti126. Epub 2005 Oct 12. PMID 16221917
- [Result] Gary TL, Batts-Turner M, Bone LR, Yeh HC, Wang NY, Hill-Briggs F, Levine DM, Powe NR, Hill MN, Saudek C, McGuire M, Brancati FL. A randomized controlled trial of the effects of nurse case manager and community health worker team interventions in urban African-Americans with type 2 diabetes. Control Clin Trials. 2004 Feb;25(1):53-66. doi: 10.1016/j.cct.2003.10.010. PMID 14980748
- [Derived] Gary TL, Batts-Turner M, Yeh HC, Hill-Briggs F, Bone LR, Wang NY, Levine DM, Powe NR, Saudek CD, Hill MN, McGuire M, Brancati FL. The effects of a nurse case manager and a community health worker team on diabetic control, emergency department visits, and hospitalizations among urban African Americans with type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2009 Oct 26;169(19):1788-94. doi: 10.1001/archinternmed.2009.338. PMID 19858437